CLINICAL TRIAL: NCT04497363
Title: Open Label Study for the Use of Transcranial Ultrasound Treatment of Attention Deficit Hyperactive Disorder
Brief Title: Focused Ultrasound for the Treatment of ADHD Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fUS_ADHD
Record Dates: First submitted 2020-07-22; First posted 2020-08-04 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Focused Ultrasound (Experimental): On the day of the ultrasound appointment, patients will undergo ten minutes of ultrasound targeting the anterior cingulate. The DWL Doppler ultrasound device enables visual and auditory waveform confirmation of the anterior cerebral artery, and optical tracking technology (e.g., AntNeuro Visor2™ system) may be used in tandem with the Brainsonix ultrasound device to track a patient's brain in virtual space as well as their physical location, thereby ensuring accurate placement.
  Interventions: Device: Brainsonix Pulsar 1002

INTERVENTIONS:
Device: Brainsonix Pulsar 1002 — Each participant will undergo 8 consecutive weekly sessions (each session is 10 minutes long) of focused ultrasound with the Brainsonix Pulsar 1002 device.

SUMMARY:
The purpose of this open label study is to evaluate longer term tolerability and potential effectiveness of transcranial ultrasound in people with attention deficit hyperactive disorder (ADHD).

DETAILED DESCRIPTION:
The primary cortical regions thought to be implicated in ADHD include the prefrontal, orbitofrontal, and anterior cingulate cortices. A possible treatment approach for ADHD would employ a process designed to promote healthier function of the anterior cingulate region. The anterior cingulate in particular appears to be implicated in the activation of cognitive control networks, and has been posited as an area of interest for therapeutic research on ADHD. The subjects in this research study will be recruited through medical practice and enrolled in an 8-week protocol to undergo 8 consecutive weekly ultrasound sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Attention Deficit Hyperactive Disorder (ADHD)
* Failure to respond to traditional symptom management (e.g. stimulants, psychoeducation, cognitive-behavior therapy, etc.)
* Score of at least 8 (4 ADHD-positive items) on the Adult ADHD Self-Report Questionnaire (ASRS-V1.1)
* At least 18 years of age

Exclusion Criteria:

* • Subjects unable to give informed consent

  * Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
  * Recent surgery or dental work within 3 months of the scheduled procedure.
  * Pregnancy, women who may become pregnant or are breastfeeding
  * Advanced terminal illness
  * Any active cancer or chemotherapy
  * Any other neoplastic illness or illness characterized by neovascularity
  * Macular degeneration
  * Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
  * Advanced kidney, pulmonary, cardiac or liver failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS-v1.1) | Baseline
  This instrument is designed to evaluate for severity of symptoms as specified in the DSM-IV-TR. The ASRS is composed of 18 questions, and uses a scale that ranges from 0-4 based on the individuals mark in either the "never, rarely, sometimes, often, very often" column for a possible total score of 72. The minimum score to qualify for study inclusion is 8 (i.e., 4 or more "symptom-positive" answers), and the maximum possible score is 72. The higher the score, the more indicative of higher severity of ADHD symptoms. Each column is used to describe the severity of the individuals symptoms based on the questions asked. Each participant is asked to make a mark within one column for each question that best describes their answer. The first 6 questions of the scale comprise Part A, which is more generally used as a screening measure. Questions 12-18 comprise Part B, which provides further identifying clues for individual symptoms.

SECONDARY OUTCOMES:
Adult ADHD Self-Report Scale (ASRS-v1.1) | Post Final Treatment (8 weeks from baseline)
  This instrument is designed to evaluate for severity of symptoms as specified in the DSM-IV-TR. The ASRS is composed of 18 questions, and uses a scale that ranges from 0-4 based on the individuals mark in either the "never, rarely, sometimes, often, very often" column for a possible total score of 72. The higher the score, the more indicative of higher severity of ADHD symptoms. Each column is used to describe the severity of the individuals symptoms based on the questions asked. Each participant is asked to make a mark within one column for each question that best describes their answer. The first 6 questions of the scale comprise Part A, which is more generally used as a screening measure. Questions 12-18 comprise Part B, which provides further identifying clues for individual symptoms. Improvement will be gauged by reduction in overall score (minimally clinically important difference will be 20% for this study).

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates of West Los Angeles
Locations (2):
- United States (2):
  - Neurological Associates of West LA, Santa Monica, California
  - Neurological Associates of West Los Angele, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- [Background] Coupe P, Manjon JV, Lanuza E, Catheline G. Lifespan Changes of the Human Brain In Alzheimer's Disease. Sci Rep. 2019 Mar 8;9(1):3998. doi: 10.1038/s41598-019-39809-8. PMID 30850617
- [Background] Drevets WC, Savitz J, Trimble M. The subgenual anterior cingulate cortex in mood disorders. CNS Spectr. 2008 Aug;13(8):663-81. doi: 10.1017/s1092852900013754. PMID 18704022
- [Background] Mayberg HS, Brannan SK, Mahurin RK, Jerabek PA, Brickman JS, Tekell JL, Silva JA, McGinnis S, Glass TG, Martin CC, Fox PT. Cingulate function in depression: a potential predictor of treatment response. Neuroreport. 1997 Mar 3;8(4):1057-61. doi: 10.1097/00001756-199703030-00048. PMID 9141092
- [Background] Chan E, Fogler JM, Hammerness PG. Treatment of Attention-Deficit/Hyperactivity Disorder in Adolescents: A Systematic Review. JAMA. 2016 May 10;315(18):1997-2008. doi: 10.1001/jama.2016.5453. PMID 27163988
- [Background] Dunn GA, Nigg JT, Sullivan EL. Neuroinflammation as a risk factor for attention deficit hyperactivity disorder. Pharmacol Biochem Behav. 2019 Jul;182:22-34. doi: 10.1016/j.pbb.2019.05.005. Epub 2019 May 16. PMID 31103523
- [Background] Amico F, Stauber J, Koutsouleris N, Frodl T. Anterior cingulate cortex gray matter abnormalities in adults with attention deficit hyperactivity disorder: a voxel-based morphometry study. Psychiatry Res. 2011 Jan 30;191(1):31-5. doi: 10.1016/j.pscychresns.2010.08.011. Epub 2010 Dec 3. PMID 21129938
- [Background] Shaw P, Malek M, Watson B, Greenstein D, de Rossi P, Sharp W. Trajectories of cerebral cortical development in childhood and adolescence and adult attention-deficit/hyperactivity disorder. Biol Psychiatry. 2013 Oct 15;74(8):599-606. doi: 10.1016/j.biopsych.2013.04.007. Epub 2013 May 28. PMID 23726514
- [Background] Arnsten AF, Rubia K. Neurobiological circuits regulating attention, cognitive control, motivation, and emotion: disruptions in neurodevelopmental psychiatric disorders. J Am Acad Child Adolesc Psychiatry. 2012 Apr;51(4):356-67. doi: 10.1016/j.jaac.2012.01.008. Epub 2012 Mar 3. PMID 22449642
- [Background] Materna L, Wiesner CD, Shushakova A, Trieloff J, Weber N, Engell A, Schubotz RI, Bauer J, Pedersen A, Ohrmann P. Adult patients with ADHD differ from healthy controls in implicit, but not explicit, emotion regulation. J Psychiatry Neurosci. 2019 Sep 1;44(5):340-349. doi: 10.1503/jpn.180139. PMID 31025560
- [Background] Tang C, Wei Y, Zhao J, Nie J. Different Developmental Pattern of Brain Activities in ADHD: A Study of Resting-State fMRI. Dev Neurosci. 2018;40(3):246-257. doi: 10.1159/000490289. Epub 2018 Jul 13. PMID 30153660